CLINICAL TRIAL: NCT05895331
Title: The Effects of Dexmedetomidine on Thiol/Disulphide Homeostasis in Coronary Bypass Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Özgüner, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: AnkaraEtlikYusufOzguner001
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Dexmedetomidine; Oxidative Stress
Keywords: Disulphide; Thiol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dexmedetomidine used group in Coronary Bypass Surgery
  Interventions: Diagnostic Test: Thiol/Disulphide Homeostasis
- Dexmedetomidine non-used group in Coronary Bypass Surgery
  Interventions: Diagnostic Test: Thiol/Disulphide Homeostasis

INTERVENTIONS:
Diagnostic Test: Thiol/Disulphide Homeostasis — An automated analysis quantitatively measuring serum native and total thiol, and disulfides has been recently described as a method to determine dynamic Thiol/Disulfide Homeostasis (TDH).

SUMMARY:
Dexmedetomidine (DEX) is a sedative and anesthetic drug with known antioxidant properties.In this study, it was aimed to investigate the oxidative stress levels in patients undergoing on-pump CABG by measuring the thiol/disulfide levels and to investigate the effects of dexmedetomidine infusion used in Coronary Bypass Surgery on dynamic Thiol/Disulphide Homeostasis.

DETAILED DESCRIPTION:
It is well known that cardiovascular disease is the leading cause of increased morbidity and mortality worldwide. One of the key surgical procedures that patients with coronary artery disease (CAD) are often subjected to is coronary artery bypass grafting (CABG). However, the cardiopulmonary bypass (CPB) pump increases systemic oxidative stress . High levels of molecular oxygen enter the body during cardiopulmonary bypass (CPB) and reperfusion, followed by inflammation leading to the formation of free oxygen radicals which causes lipid peroxidation, ultimately resulting in an oxidative attack at the cell and tissue level.

Thiols are organic sulphur derivatives containing Sulfhydryl Residues (-SH) in their active regions. Thiols easily react with oxygen containing free radicals to form disulfides. This is a defence mechanism against oxidative stress.7 An automated analysis quantitatively measuring serum native and total thiol, and disulfides has been recently described as a method to determine dynamic Thiol/Disulfide Homeostasis (TDH).The role of dynamic thioldisulfide homeostasis has been increasingly shown in many diseases. There is a growing number of evidences that an abnormal thiol-disulfide homeostasis may play role in the pathogenesis of a variety of diseases such as cardiovascular disease, malignancies, rheumatoid arthritis, chronic kidney disease, and acquired immunodeficiency syndrome.

Dexmedetomidine (DEX) is a sedative and anesthetic drug with known antioxidant properties.In this study, it was aimed to investigate the oxidative stress levels in patients undergoing on-pump CABG by measuring the thiol/disulfide levels and to investigate the effects of dexmedetomidine infusion used in Coronary Bypass Surgery on dynamic Thiol/Disulphide Homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone coronary bypass surgery using a cardiopulmonary pump
* Patients who agreed to participate in the study

Exclusion Criteria:

* Bypass surgeries without cardiopulmonary pump
* Patients with intraoperative unexpected/undesirable complications
* Patients who did not agree to participate in the study
* Patients with missing data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone coronary bypass surgery using a cardiopulmonary pump
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-05 (Estimated); Primary Completion 2023-09-05 (Estimated); Study Completion 2023-10-05 (Estimated)

PRIMARY OUTCOMES:
Thiol/Disulphide Homeostasis | 30 min before the start of surgery
  An automated analysis quantitatively measuring serum native and total thiol, and disulfides has been recently described as a method to determine dynamic Thiol/Disulfide Homeostasis (TDH).
Thiol/Disulphide Homeostasis | at the time of aortic cross clamp off
  An automated analysis quantitatively measuring serum native and total thiol, and disulfides has been recently described as a method to determine dynamic Thiol/Disulfide Homeostasis (TDH).
Thiol/Disulphide Homeostasis | at the time of surgery over
  An automated analysis quantitatively measuring serum native and total thiol, and disulfides has been recently described as a method to determine dynamic Thiol/Disulfide Homeostasis (TDH).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Varlık Mahallesi, Halil Sezai Erkut Caddesi Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erel O, Neselioglu S. A novel and automated assay for thiol/disulphide homeostasis. Clin Biochem. 2014 Dec;47(18):326-32. doi: 10.1016/j.clinbiochem.2014.09.026. Epub 2014 Oct 7. PMID 25304913
- [Background] Akkus O, Kaypakli O, Koca H, Topuz M, Kaplan M, Baykan AO, Samsa MZ, Quisi A, Erel O, Neselioglu S, Gur M. Thiol/disulphide homeostasis in thoracic aortic aneurysm and acute aortic syndrome. Biomark Med. 2018 Apr;12(4):349-358. doi: 10.2217/bmm-2017-0372. Epub 2018 Feb 13. PMID 29436236
- [Background] Vukicevic P, Klisic A, Neskovic V, Babic L, Mikic A, Bogavac-Stanojevic N, Matkovic M, Milicevic V, Aleksic N, Kotur-Stevuljevic J. Oxidative Stress in Patients before and after On-Pump and Off-Pump Coronary Artery Bypass Grafting: Relationship with Syntax Score. Oxid Med Cell Longev. 2021 Jul 30;2021:3315951. doi: 10.1155/2021/3315951. eCollection 2021. PMID 34381560
- [Background] Unchiti K, Leurcharusmee P, Samerchua A, Pipanmekaporn T, Chattipakorn N, Chattipakorn SC. The potential role of dexmedetomidine on neuroprotection and its possible mechanisms: Evidence from in vitro and in vivo studies. Eur J Neurosci. 2021 Nov;54(9):7006-7047. doi: 10.1111/ejn.15474. Epub 2021 Oct 25. PMID 34561931
- [Derived] Ozguner Y, Altinsoy S, Kulturoglu G, Unal D, Ergil J, Neselioglu S, Erel O. The effects of dexmedetomidine on thiol/disulphide homeostasis in coronary artery bypass surgery: a randomized controlled trial. BMC Anesthesiol. 2024 Nov 7;24(1):402. doi: 10.1186/s12871-024-02794-1. PMID 39511476